CLINICAL TRIAL: NCT04466163
Title: Strengthening the Healthy Adult Mode: a Case Experimental Study Exploring the Effects of a New Schema Therapy Protocol in an Adult Outpatient Population
Acronym: ST-HA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, Yvonne Versluis, Healthcare Psychologist, Clinical Psychologist in training, Zuyderland Medisch Centrum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST-HA
Record Dates: First submitted 2020-06-29; First posted 2020-07-10 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Trauma, Psychological; Personality Disorders; Chronic Psychiatric Disorder
Keywords: Schema Therapy; Positive Psychology; Self-compassion; Personality disorder; Well-being; Positive Affect; Healthy Adult mode
MeSH Terms: conditions — Psychological Trauma; Personality Disorders | interventions — Schema Therapy

STUDY DESIGN:
Intervention Model Description: In this study a single case experimental design (n = 8) with multiple measures will be used, to determine the effects of the ST-HA protocol on self-compassion, well-being, positive affect and Healthy Adult functioning. For each participant a no-treatment randomized baseline period (2-5 weeks) will be compared with treatment (ST-HA, 10 weekly sessions) and post-treatment follow-up (at 1- and 3-months).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schema Therapy and the Healthy Adult (Experimental): For this study the ST-HA protocol outlined by Broersen & Claassen (2019) will be followed, consisting of ten one-and-a-half hour individual sessions across ten weeks with daily homework assignments (30-60 minutes). The ST-HA protocol is based on three pillars, aimed at improving self-compassion, well-being and positive affect. First psycho-education about compassionate affect regulation is given and patients learn to recognize the importance of self-caring behavior in stimulating the soothing- affect system to buffer against stress. The second pillar of the ST-HA protocol concerns the development of personal values and committed action as well as getting insight in values of important others. The third pillar concerns developing self-compassion
  Interventions: Behavioral: Schema Therapy and the Healthy Adult
- Baseline (No Intervention): Outcome variables will be measured repeatedly in a pre-treatment baseline condition (2-5 weeks). Patients are randomly assigned to a pre-treatment/baseline phase. In the present study a restricted randomisation is chosen (Heyvaert & Onghena, 2014a). A minimum length of the phases is decided a priori in order to prevent for the assignment of too few measurements per phase and to ensure that the full treatment protocol can be offered

INTERVENTIONS:
Behavioral: Schema Therapy and the Healthy Adult — The protocol 'Schematherapy and the Healthy Adult' (ST-HA, Broersen & Claassen, 2019) is a direct intervention meant to strengthen patients' healthy adult functioning by developing compassion and care for well-being in the face of (childhood) adversity.
  Arms: Schema Therapy and the Healthy Adult

SUMMARY:
Background: Strengthening the Healthy Adult schema mode is the ultimate goal in Schema Therapy, working as an assumed mechanism of long-term change through improved positive mental health. Evidence-based interventions to directly strengthen this Healthy Adult mode are sparse.

Objective: To study the feasibility, acceptability and effectiveness of the treatment protocol 'Schema Therapy and the Healthy Adult' (ST-HA) during the final stage of schema therapy in adult outpatients with personality- or chronic psychopathology. Method: In this study a single case experimental design (n = 8) with multiple measures will be used, to determine the effects of the ST-HA protocol on self-compassion, well-being, positive affect and Healthy Adult functioning. For each participant a no-treatment randomized baseline period (2-5 weeks) will be compared with treatment (ST-HA, 10 weekly sessions) and post-treatment follow-up (at 1- and 3-months). Assessments include brief diaries regarding self-compassion and Healthy Adult functioning (daily from baseline to end of intervention, and 7-days at 1- and 3-months follow-up) and standardized questionnaires for measuring weekly changes in self-compassion, well-being and adaptive schema modes. During phase changes additional measures of trait self-compassion, positive affect, adaptive schema modes and symptomatic distress will be administered.

DETAILED DESCRIPTION:
Schema therapy (ST; Young, 1990, Young et al., 2003) is an effective treatment for personality disorders and other chronic psychopathology, leading to significant improvement in functioning in most patients. The model of psychopathology that underlies ST is based on the assumption that when core emotional needs - especially those related to attachment stability - are insufficiently met in childhood, there is an increased chance that long-standing patterns of maladaptive thinking, feeling, behaving and coping (called schemas) will develop (i.e. Hawke & Provencher, 2011; Flink et al., 2019; Lockwood & Peris, 2012). When schemas are activated, the individual switches into a specific emotional-cognitive-behavioral state, called schema mode.

Schema therapy formulated in mode terms aims to build a Healthy Adult mode in patients by correcting dysfunctional self-representations which originate from unmet childhood needs (child modes), thereby replacing internalized critic modes with adaptive coping behavior (e.g. Arntz & Jacob, 2012; Claassen & Pol, 2013, 2014; Lobbestael et al., 2007; Young et al., 2003). This healthy, adultlike part of the self helps patients to meet their emotional needs and seems related to a longer-term view of emotional well-being (Roediger, Stevens, & Brockman, 2018). Recent studies demonstrate that building the Healthy Adult mode is crucial for long-term outcomes in patients with schema-driven perception and behavior, working as a mechanism of change through improved positive emotion regulation strategies to cope with (childhood) adversity (Louis et al., 2018; Westerhof & Wolterink, 2018; Yakin et al., 2020). A more explicit focus on healthy emotional functioning and regulation within ST seems therefore important. One useful emotional-approach coping strategy associated with healthy adult functioning is self-compassion (Trompetter et al., 2016; Yakin et al., 2019). Self-compassion is defined as being kind toward oneself (Neff, 2003b) and being able to use self-reassurance and soothing when presented with negative affect or adversities (Gilbert, 2010; Gilbert et al., 2017; Kirschner et al. 2019). It is facilitated by early experiences of care and warmth from an attachment ﬁgure, which contributed to a sense of safeness in which individuals develop a soothing-affective system (Brophy et al., 2020; Gilbert, 2014; Gilbert & Proctor, 2006; Mackintosh et al., 2018). This system exerts its protective function by stimulating physiological processes associated with stress reduction and positive affiliation affects (i.e. feeling loved, safe and securely attached) (Depue & Morrone-Strupinsky, 2005; Engen & Singer, 2015; Porges, 2007). Promoting the soothing-affective system subsequently helps reducing threat-related negative emotional states and excessive drive-related arousal (i.e. activation of dysfunctional schema modes) by increasing compassionate self-reassuring abilities, which are characterized by a caring, warm, and accepting attitude toward the self (Gilbert, 2010; Petrocchi et al., 2019; Thimm, 2017). Self-compassion therefore increases positive self, while reducing negative self (Mackintosch et al., 2018; Kirschner et al. 2019) via addressing dysfunctional schema modes. That is, the healthy side of patients is aware of self-undermining messages, can challenge them, hereby reducing their impact by practicing self-compassion with focus on attunement to emotional needs. Self-compassion and the ability to cultivate positive emotions in ourselves can thus be viewed as strategy to 'broaden- and build' healthy adult behavior (Fredrickson, 2001). Positive emotions allow us to discard habitual modes and instead look for flexible, new ways of thinking and acting (Fredrickson, 2003, 2004; Fredrickson et al., 2008). This broadened mindset can accumulate and compound to build biological (e.g. cardiac vagal tone) as well as cognitive (e.g. mindfulness), social (e.g. positive relations) and psychological (e.g. life-purpose) resources (Cloninger, 2006; Cloninger & Zohar, 2011). Experiencing positive emotions subsequently increases functional coping in a needs-based, value-driven, flexible way, serving as 'compass' for healthy adult behavior over lifetime (Bahner, 2016; Deci & Ryan, 2000; Plumb et al., 2009; Schreurs & Westerhof, 2013).

Against this background, interventions focusing on the integration of schema therapy and compassion based therapy seems promising. To our best knowledge the protocol 'Schematherapy and the Healthy Adult' (ST-HA, Broersen & Claassen, 2019) is the first direct intervention meant to strengthen patients' healthy adult functioning by developing compassion and care for well-being in the face of (childhood) adversity. The current study explores the effectiveness, acceptability and feasibility of the ST-HA protocol in adult outpatients with personality- or chronic psychopathology during final stage ST, in which there is a focus on positive mental health, resilience and preparing therapy termination. It is hypothesized that administering the ST-HA protocol: (1) will increase self-compassion, well-being, positive affect and adaptive schema modes over the intervention and follow-up period, measured by daily diary data and standardized measurements; (2) will be accompanied by self-reported symptom-reduction over the intervention and follow-up period; and (3) will be acceptable and feasible in adult outpatients.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 to 65 year
* a diagnosis of personality disorder and/or (comorbid) persistent mood-/somatic symptom disorder according to DSM-5 at the start of regular group or individual ST;
* following final stage individual or group ST (as indicated by the patients' certified Schema Therapist). If ST is terminated, this must be within four months before starting with current ST-HA study;
* suboptimal positive mental health as indicated by low to moderate levels of well-being, determined by the Mental Health Continuum
* Short Form (MHC-SF; Keyes, 2002; Lamers et al., 2011) or below average to low scores on the Positive Affect scale of the Positive And Negative Affect Schedule (PANAS; Watson et al., 1988);
* self-reported motivation for a 10-session psychological intervention focusing on positive mental health;
* have access to a computer or tablet with a good Internet connection;
* possess an e-mail address;
* have sufficient proficiency of the Dutch language (reading and writing);
* provided informed consent.

Exclusion Criteria:

* severe psychiatric disorders: acute suicidal risk, a psychotic and/or bipolar disorder, schizophrenia, delirium, dementia of severe cognitive impairment;
* ongoing other ST/psychological treatment during the baseline and treatment phase;
* former treatment based on the ST-HA protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Diary: Healthy Adult Functioning change | daily during baseline (14-35 days) and intervention (10 weeks), one week after 1 month/3 months
  To check change in self-reported self-compassion a diary will be used consisting of a subset of seven items measuring compassionate affect, reasoning and behavior selected from standardized questionnaires with visual analog scales (VAS) (Morley, 2017; see: Vlaeyen et al., 2001). Five items adapted from the Safe/Content Affect Scale (Gilbert et al., 2008), will ask patients about their soothing affiliative affect (i.e. feeling safe, secure, content, warm). Two items ask patients about state self-reassuring and -kindness and are adopted from the Self-Compassion Scale (SCS; Neff, 2003a; see Kirschner et al., 2019). The three last diary items represent patient-generated goals, referring to personally relevant self-caring and supportive Healthy Adult behaviors. These personalized items can include healthy attitudes, choices, preferences and opportunities, that patients are willing to engage in.
State Self-Compassion (Change) | weekly during baseline (14-35 days) & intervention period (10 weeks), 1 month follow-up, 3 month follow-up
  State self-compassion will be measured by the State Self-Compassion Scale - Short Form (SSCS-SF; Neff et al., submitted). Participants are instructed to think about a situation that they are experiencing right now, that is painful or difficult. Participants subsequently have to indicate how well each of six statements applies to how they are feeling toward themselves right now as they think about this situation on a five point scale, ranging from 1 ('not at all true for me') to 5 ('very true for me'). The SSCS-SF is a valid and reliable measure of state self-compassion (Neff et al., submitted).
Trait Self-Compassion (Change) | weekly during baseline (14-35 days) & intervention period (10 weeks), 1 month follow-up, 3 month follow-up
  Trait self-compassion will be measured by the 12-item short form of the Self-Compassion Scale (SCS-SF; Raes et al., 2010).
Self-Criticism and Self-Reassuring (Change) | weekly during baseline (14-35 days) & intervention period (10 weeks), 1 month follow-up, 3 month follow-up
  Self-criticism and self-reassurance and will be measured by the Forms of Self-Criticism/-Reassurance Subscales- Short form (FSCRS-SF; Sommers-Spijkerman et al., 2018).
Well-being (Change) | weekly during baseline (14-35 days) & intervention period (10 weeks), 1 month follow-up, 3 month follow-up
  Well-being will be measured by the Mental Health Continuum-Short Form (MHC-SF; Lamers et al., 2011), a 14-item self-report questionnaire covering three core components of well-being: (1) emotional wellbeing, deﬁned in terms of positive feelings (e.g. happiness and positive affect) and satisfaction with life (three items); (2) psychological wellbeing; deﬁned in terms of positive functioning in individual life (e.g. feelings of self-acceptance, environmental mastery, purpose in life, positive social relationships) (six items) and (3) social wellbeing, deﬁned in terms of positive functioning in community life (e.g. feelings of social contribution, social acceptance, and social integration) (ﬁve items).
Schema Modes (Change) | SMI: start baseline (week 0), start intervention (after 14-35 days of baseline), after 10 weeks of intervention, 1 month follow-up, 3 month follow-up.
  Adaptive schema modes will be measured with the Schema Modi Inventory (SMI; Young et al., 2007).
Positive Affect (Change) | weekly during baseline (14-35 days) & intervention period (10 weeks), 1 month follow-up, 3 month follow-up
  Positive affect will be measured by the Positive Affect Subscale (PA) of the PANAS (Watson et al., 1988).
Momentary Schema Mode Inventory (Change) | Momentary SMI: weekly during baseline (up to 14-35 days) & intervention period (10 weeks), 1 month follow-up, 3 month follow-up
  Also, the Momentary Schema Mode Inventory, adapted from the SMI for weekly assessment of modes (Roelofs et al., 2016) will be used.

SECONDARY OUTCOMES:
Symptomatic distress (Change) | 5 timepoints (start baseline (week 0), start intervention (after 14-35 days of baseline), after 10 weeks of intervention, 1 month follow-up, 3 months follow-up
  Symptomatic distress will be measured by the Outcome Questionnaire-45 (OQ-45; De Jong et al., 2007; Lambert et al., 2004).

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland MC, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: Jan. 2022 (6 months)